CLINICAL TRIAL: NCT06338683
Title: Survival With the Addition of Olanzapine to Anticancer Therapy in Patients With Locally Advanced, Unresectable or Metastatic Gastric, Esophageal, Hepatopancreaticobiliary and Lung Cancer: a Randomized Clinical Trial
Brief Title: Survival With Olanzapine in Patients With Locally Advanced or Metastatic Upper Gastrointestinal and Lung Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qinghai Red Cross Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QRCH-2024001
Record Dates: First submitted 2024-03-21; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Advanced Cancer; Olanzapine; Progression Free Survival
Keywords: advanced cancer; olanzapine; chemotherapy; progression free survival
MeSH Terms: interventions — Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (ONS group) (Experimental): Patients receive olanzapine 2.5mg PO until disease progression. Intervention: Patients received olanzapine and nutritional advice and standard antitumor treatment.
  Interventions: Drug: Olanzapine 2.5 MG; Drug: Standard anti-tumor treatment; Dietary Supplement: Nutritional advice
- Arm II (NS group) (Placebo Comparator): No Intervention: Patients received nutritional advice and standard anti-tumor treatment.
  Interventions: Drug: Standard anti-tumor treatment; Dietary Supplement: Nutritional advice

INTERVENTIONS:
Drug: Olanzapine 2.5 MG — Oral olanzapine 2.5 mg once daily at bedtime until disease progression
  Arms: Arm I (ONS group)
Drug: Standard anti-tumor treatment — Clinicians choose the appropriate standard antitumor drug therapy based on the patient's specific situation
Dietary Supplement: Nutritional advice — All patients enrolled in the study were required to undergo a nutritional assessment and were provided with nutritional advice based on their condition

SUMMARY:
This study aims to assess the impact of adding olanzapine to nutritional advice and standard anti-tumor therapy on the survival and safety of patients with locally advanced, unresectable or metastatic gastric cancer, esophageal cancer, hepato-pancreaticobiliary cancer, and lung cancer. Researchers seek to determine whether olanzapine can improve progression-free survival (PFS), overall survival (OS), and objective response rate (ORR) in advanced cancer patients who received standard anti-tumor therapy, and investigate the relationship between olanzapine-induced weight changes and patient survival.

DETAILED DESCRIPTION:
This study is a prospective, randomized, multicenter, open-label clinical trial to evaluate the effect of olanzapine on survival in patients with locally advanced, unresectable, or metastatic gastric, esophageal, hepato-pancreaticobiliary, and lung cancer. Patients who meet the inclusion and exclusion criteria will be formally enrolled after screening and signing an informed consent form. Eligible patients will be dynamically randomized in a 1:1 ratio to either the Olanzapine + Nutritional advice + Standard anti-tumor treatment group (ONS group) or the Nutritional advice + Standard anti-tumor treatment group (NS group). The ONS group will receive olanzapine treatment orally until disease progression. Survival outcomes, including median PFS, OS, and ORR, will be monitored during treatment through follow-up assessments.

In addition, baseline and post-treatment weight data will be collected to assess the incidence of weight loss and changes in body mass index (BMI) among patients. Researchers will collect survey questionnaires and conduct blood analyses to evaluate improvements in other symptoms associated with olanzapine and changes in quality of life and inflammatory markers. Primary and secondary study outcomes and adverse events will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older;
2. Eastern Cooperative Oncology Group performance status of 0-3;
3. Stage III or IV inoperable or metastatic gastric cancer, esophageal cancer, hepato-pancreaticobiliary cancer and lung cancer confirmed by histology or cytology;
4. Subjected to palliative systemic chemotherapy, regardless of first-line or second-line treatment;
5. Expected survival ≥ 3 months;
6. The patient is eligible for oral administration without dietary restrictions;
7. Exhibits a favorable adherence to treatment and follow-up, demonstrates compliance with the research protocol, and willingly signs the informed consent form.

Exclusion Criteria:

1. Weight loss and gain may be attributed to alternative factors, such as edema or ascites;
2. Suffers from mental disorders or is under the medication of any antipsychotic or antidepressant drugs;
3. History of central nervous system disorders (such as brain metastasis, epilepsy;
4. Patients undergoing sustained administration of sedative medications or long-term hormonal therapy, individuals with chronic alcoholism, or those with substance dependence on medications;
5. Prohibition of Olanzapine Intake for Contraindicated Individuals;
6. History of clozapine-induced agranulocytosis because patients will be at increased risk for neutropenia with Olanzapine;
7. Uncontrolled diabetes mellitus and Uncontrolled seizure disorder;
8. Pregnant and Nursing women;
9. Exclusion criteria include active participation in another interventional clinical trial, ongoing involvement in an observational (noninterventional) clinical trial, or being in the survival follow-up phase of an interventional clinical trial;
10. Researchers posit that any condition deemed potentially harmful to the subjects or that might prevent subjects from meeting or adhering to the research requirements shall not be permissible for inclusion in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2027-03-20 (Estimated); Study Completion 2028-03-20 (Estimated)

PRIMARY OUTCOMES:
Comparing the difference in Median PFS between the two groups | 2 years
  PFS was defined as the time between the start of treatment in this study and the onset of (any aspect of) tumor progression or death (from any cause). Assessment through the RECICT 1.1 version of solid tumors

SECONDARY OUTCOMES:
Comparing the difference in Median OS between the two groups | 2 years
  OS was defined as the time from the start of randomization to death due to any cause. Assessment through the RECICT 1.1 version of solid tumors
Comparing the difference in ORR between the two groups | 2 years
  ORR was defined as the proportion of patients with advanced disease who achieved complete or partial remission after treatment. Assessment through the RECICT 1.1 version of solid tumors
Comparing the difference in the incidence of ≥3% weight loss between the two groups | 2 years
  Patients will receive weight measurements every 2 cycles. Over a 2-year period, the incidence of ≥3% weight loss until progression between the two groups will be assessed based on patients' baseline and post-treatment measurements to determine the efficacy of the drug.
Comparing the difference in BMI between the two groups | 2 years
  The BMI will be calculated by dividing weight in Kg with the square of the body height (in m2), and is expressed in units of kg/m2. Weight will be recorded by a high quality calibrated digital scale. Participants would be instructed to keep light cloths according to their comfort and no foot-ware. Weight will be expressed in kilograms (Kg) and same machine will be used during each recoding, preferably during the same hour of the day. Height will be measured using a stadiometer, in centimeters (cm) using the metric system. Comparison of BMI (BMI <20 kg/m2; BMI 20-25 kg/m2; BMI >25 kg/m2) between the two groups
Comparing the difference in the improvement in other symptoms (appetite, nausea, fatigue, insomnia) between the two groups | 2 years
  Patients will be asked to fill the Functional Assessment of Anorexia/Cachexia Therapy (FAACT) Anorexia/Cachexia Subscale (A/CS) questionnaire (investigator assisted) for the other symptoms both validated with a set cut-off values before start of chemotherapy treatment and after every 2 weeks. These instruments will be presented to the patients on paper and assistance will be offered if required. Both instruments will be filled out based on the patient's experience regarding their appetite during the last 7 days. The 12 items of the FAACT-A/CS are scored on a five-point Likert scale (0 = not at all, 1 = a little bit, 2 = somewhat, 3 = quite a bit, and 4 = very much). The scores of negatively worded items should be reversed. The sum score ranges from 0 to 48, whereby a lower score indicates less appetite. For scoring the FAACT-A/CS, the FACIT manual will be applied. The cut-off values of ≤37 on the FAACT-A/CS had the highest predictive values.
Comparing the difference in Quality of life in the overall stage between the two groups | 2 years
  Assessment through the EuroQol Five Dimensions Questionnaire (EQ-5D). EQ-5D is a standardized instrument used for assessing an individual's health-related quality of life. It comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has three levels that describe the person's level of functioning or well-being in that specific area. Additionally, EQ-5D includes a visual analog scale where individuals rate their overall health on a scale from 0 (worst imaginable health) to 100 (best imaginable health)
neutrophil-to-lymphocyte ratio | 2 years
  Comparing the difference in Changes in inflammatory factor neutrophil-to-lymphocyte ratio
platelet-to-lymphocyte ratio | 2 years
  Comparing the difference in Changes in inflammatory factor
C-reactive protein (CRP) concentration | 2 years
  Comparing the difference in Changes in inflammatory factor
concentration of albumin | 2 years
  Comparing the difference in Changes in inflammatory factor
Level of interleukin (IL)-6 and IL-8 | 2 years
  Comparing the difference in Changes in inflammatory factor , through the examination of blood profiles
Comparing the difference in the side effects of olanzapine treatment between the two groups | 2 years
  The proportion of side effects related to olanzapine treatment in patients evaluated by Common Terminology Criteria for adverse events Version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Qinghai Red Cross Hospital, Xining, Qinghai, China